CLINICAL TRIAL: NCT00596622
Title: Dysfunctional Cortico-Limbic Activity and Connectivity in Bipolar Disorder Before and After Lithium Treatment: An fMRI Study
Brief Title: FMRI Study of Brain Response Before and After Lithium Treatment in People With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01MH075025 (NIH); 0607-23 (Other: Indiana University IRB); DATR A3-NSS (Other: Indiana University); R01MH075025 (NIH)
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Bipolar Disorder
Keywords: Major Depressive or Manic Episodes; Bipolar; Mania; Depression; Lithium; fMRI; Pictures; Brain Scan
MeSH Terms: conditions — Bipolar Disorder; Mania; Depression | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bipolar Manic Subjects Treated (Experimental): Bipolar mania picture response during fMRI before and after treatment with lithium
  Interventions: Drug: Lithium
- Bipolar Depressed Subjects Treated (Experimental): Bipolar depression picture response during fMRI before and after treatment with lithium
  Interventions: Drug: Lithium
- Bipolar Euthymic Subjects Treated (Experimental): Bipolar euthymia picture response before and after treatment with lithium
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.

SUMMARY:
This study will assess the effects of bipolar disorder on brain activity and will determine if medication changes the brain activity in people with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic brain disorder that causes dramatic changes in a person's mood and energy. People with BD undergo periods of extreme happiness and extreme sadness, known as episodes of mania and depression. A person undergoing an episode of mania often experiences euphoric moods, increased energy, and aggressive behaviors, while a person in a depressed state often experiences low moods, lack of energy, and feelings of sadness. Researchers have recently discovered that abnormalities in certain brain areas that control emotion are often present in those with BD. It is believed that the severe mood shifts in BD may cause alterations in normal brain activity, specifically in corticolimbic activation and connectivity. Current mood stabilizing medications used to treat people with BD may help normalize these brain activity abnormalities. This study will assess the effects of BD on brain activity using functional magnetic resonance imaging (fMRI) and will determine if treatment with lithium changes the brain activity in people with BD.

This 9-week study will include participants who are healthy, have BD, or are siblings of subject with BD. All potential participants will undergo initial testing, which will include a physical examination, blood tests, and an electrocardiogram (EKG). Participants will also be asked to answer questions about their mental health, drug use, personality, family history, and psychological well-being. Eligible participants will then return on a different day to undergo an MRI scan, taking 4 hours to complete. During the scan, participants will be asked to perform tasks designed to show changes in blood flow in specific brain regions. These tasks will include listening to sounds and looking at various letters, words, and pictures. This will mark the completion of the study for healthy participants, first degree relatives, and those participants with BD who do not wish to receive medication treatment.

Following the first MRI scan, participants with BD who wish to undergo medication treatment will begin an 8-week course of lithium. Participants will be asked to come to the clinic at least once a week for medication monitoring visits. During these visits, participants will undergo blood draws and assessments on depression and mania. Participants will return for two repeat MRI scans after Weeks 2 and 8 of lithium treatment.

ELIGIBILITY:
Inclusion criteria for BD participants:

* Meets DSM-IV criteria for bipolar I or II disorder
* Meets criteria to undergo an MRI scan based on MRI screening questionnaire
* Suited for outpatient care during the study as ascertained by a score of less than 5 on the Clinical Global Severity Scale, no significant suicidal or homicidal ideation, and no severe disability

Inclusion criteria for BD depressed participants:

* Meets criteria for DSM-IV depressive episode-current
* Score of greater than 15 but less than 30 on the 17-item HDRS
* Score of less than 12 on the Young Mania Rating Scale

Inclusion criteria for BD (hypo) manic participants:

* Meets criteria for DSM-IV manic episode-current
* Score of less than or equal to 18 on the 17-item HDRS
* Score of greater than 12 but less than 25 on the Young Mania Rating Scale

Inclusion criteria for BD euthymic patients:

* Satisfy criteria for DSM-IV for euthymic state-current for at least 2 weeks.
* 17-item Hamilton Depression Rating Scale < 12; Young Mania Rating Scale score < 10

Exclusion criteria for BD participants:

* Meets DSM-IV criteria for unipolar depression, schizophrenia, schizophreniform disorder, schizoaffective disorder, atypical psychosis, anxiety disorder as a primary diagnosis, mental retardation, or personality disorder
* Received electroconvulsive therapy in the 12 months prior to study entry
* Use of neuroleptics, mood stabilizers, or benzodiazepines in the 2 weeks prior to study entry
* Use of antidepressants in the 2 weeks prior to study entry
* Use of fluoxetine in the 5 weeks prior to study entry
* Use of lithium in the 6 months prior to study entry
* Acutely suicidal or homicidal or requiring inpatient treatment
* Meets DSM-IV criteria for substance/alcohol dependence, excluding caffeine or nicotine, in the 6 months prior to study entry or substance/alcohol abuse in the 3 months prior to study entry
* Use of alcohol in the 1 week prior to study entry and refusal to avoid alcohol use during the course of the study
* Presence of serious acute or chronic medical or neurological illness, including previously known HIV positive status (due to possible CNS involvement) as assessed by history, physical examination, and laboratory examination
* Pregnant or breastfeeding
* Metallic implants or other contraindication to MRI

Inclusion criteria for first degree relatives of bipolar disorder subjects:

* Ages 15-60 years (inclusive) and able to give voluntary informed consent.
* Have never satisfied criteria for DSM-IV BD.
* Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire.
* 17-item Hamilton Depression Rating Scale < 10; Young Mania Rating Scale score < 10

Exclusion criteria for first degree relatives of bipolar disorder subjects:

* Under 15 years of age.
* Meeting DSM-IV criteria for current episode of unipolar depression
* Pregnant or breast feeding.
* Metallic implants or other contraindication to MRI.
* Currently taking any prescription or centrally acting medications.
* Serious acute or chronic medical or neurological illness as assessed by history, physical examination and laboratory examination including CBC and blood chemistry.
* Use of alcohol in the past 1 week and not being able to avoid alcohol use during the course of the study.

Inclusion criteria for healthy subjects:

* Ages 18-60 years (inclusive) and able to give voluntary informed consent.
* No current or past history of psychiatric illness or substance abuse or dependence.
* No current or past history of psychiatric illness or substance abuse or dependence in a first degree relative.

Exclusion criteria for healthy participants:

* Under 18 years of age
* Pregnant or breastfeeding
* Metallic implants or other contraindication to MRI
* Significant family history of psychiatric or neurological illness
* Currently taking any prescription or centrally acting medications
* Serious acute or chronic medical or neurological illness as assessed by history, physical examination, and laboratory examination
* Use of alcohol in the 1 week prior to study entry and refusal to avoid alcohol use during the course of the study

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2007-08; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Psychiatric Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bipolar Subjects Who Were Included in Lithium Treatment Arm: Participants with bipolar disorder who undergo fMRI and lithium treatment
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Picture response during fMRI: While undergoing an fMRI scan, participants will be presented with pictures, letters, words, and sounds to evoke emotional responses. There will be a maximum of three MRI scans over 9 weeks.
Period: Overall Study
Arm/Group | Bipolar Subjects Who Were Included in Lithium Treatment Arm
Started | 46
Completed | 33
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- Bipolar Depressed Subjects Treated With Lithium: Participants with bipolar depression picture response during fMRI before and after treatment with lithium
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Depression and mania scores before and after treatment
- Bipolar Manic Subjects Treated With Lithium; Bipolar Euthymic Subjects Treated With Lithium: Participants with bipolar mania picture response during fMRI before and after treatment with lithium
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Depression and mania scores before and after treatment
- Total: Total of all reporting groups
Arm/Group | Bipolar Depressed Subjects Treated With Lithium | Bipolar Manic Subjects Treated With Lithium | Bipolar Euthymic Subjects Treated With Lithium | Total
Number analyzed (Participants) | 18 | 22 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10) | 34 (11) | 26 (4) | 33 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 3 | 26
  Male | 10 | 7 | 3 | 20
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 6 | 46

OUTCOME MEASURES:

1. Primary Outcome: 17-item Hamilton Depression Rating Scale (HDRS)
Description: 17-item HDRS is gold standard for measurement of depression with a range from 0 - 52. 10 - 14: mild depression; 14-20 moderate depression; >20: severe and very severe depression.
Time Frame: Measured at Baseline and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bipolar Depressed Participants Treated: Participants with bipolar depression who undergo fMRI and lithium treatment
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Picture response during fMRI: While undergoing an fMRI scan, participants will be presented with pictures, letters, words, and sounds to evoke emotional responses. There will be a maximum of three MRI scans over 9 weeks.
- Bipolar Manic Subjects Treated: Participants with bipolar mania who undergo fMRI and lithium treatment
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Picture response during fMRI: While undergoing an fMRI scan, participants will be presented with pictures, letters, words, and sounds to evoke emotional responses. There will be a maximum of three MRI scans over 9 weeks
- Bipolar Euthymic Subjects Treated: Participants with bipolar euthymia who undergo fMRI and lithium treatment
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Picture response during fMRI: While undergoing an fMRI scan, participants will be presented with pictures, letters, words, and sounds to evoke emotional responses. There will be a maximum of three MRI scans over 9 weeks
Arm/Group | Bipolar Depressed Participants Treated | Bipolar Manic Subjects Treated | Bipolar Euthymic Subjects Treated
Number analyzed (Participants) | 15 | 14 | 4
units on a scale
  Baseline 17-item HDRS | 20 (4) | 6 (3) | 6 (4)
  After 8 weeks lithium treatment | 2 (3) | 3 (2) | 2 (3)

2. Secondary Outcome: Young Mania Rating Scale
Description: Gold standard scale to measure mania, Range 0 - 60; 12 - 15 mild mania; 15 - 20 moderate mania; >20 severe mania
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bipolar Manic Subjects Treated | Bipolar Depressed Subjects Treated | Bipolar Euthymic Subjects Treated
Number analyzed (Participants) | 14 | 15 | 4
units on a scale
  Baseline 17-item YMRS | 15 (1) | 3 (2) | 1 (1)
  Post 8 week treatment YMRS | 3 (2) | 2 (3) | 2 (3)

ADVERSE EVENTS:
Groups:
- Bipolar Participants Treated: Participants with bipolar disorder who undergo fMRI and lithium treatment
  Lithium: Dosing will start as one 300-mg capsule per day and will be titrated up to four 300-mg capsules per day for a total of 8 weeks of treatment.
  Picture response during fMRI: While undergoing an fMRI scan, participants will be presented with pictures, letters, words, and sounds to evoke emotional responses. There will be a maximum of three MRI scans over 9 weeks.
  Adverse Events information was collected irrespective of the sub-grouping
Arm/Group | Bipolar Participants Treated
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 40/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bipolar Participants Treated (N=46)
Increased appetite (Gastrointestinal disorders) | 5
headaches (Nervous system disorders) | 15
Drymouth (Gastrointestinal disorders) | 5
blurred vision (Eye disorders) | 3
dizziness (Nervous system disorders) | 5
heart palpitations (Cardiac disorders) | 5
forgetfulness (Nervous system disorders) | 3
bad taste (Gastrointestinal disorders) | 3

LIMITATIONS AND CAVEATS:
Small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No